CLINICAL TRIAL: NCT00917059
Title: Personalized Response Indicators of SSRI Effectiveness in Major Depression
Brief Title: Personalized Indicators for Predicting Response to SSRI Treatment in Major Depression (The PRISE-MD Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Ian A. Cook, M.D., University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH085925 (NIH); R01MH085925 (NIH); 09-03-022-01; DSIR 84-CT
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Depression
Keywords: Major Depressive Disorder; SSRI; EEG
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive a 1-week treatment of escitalopram and then an 8-week treatment with escitalopram.
  Interventions: Drug: Escitalopram
- 2 (Active Comparator): Participants will receive a 1-week treatment with escitalopram and then an 8-week treatment with bupropion XL.
  Interventions: Drug: Escitalopram; Drug: Bupropion XL

INTERVENTIONS:
Drug: Escitalopram — Fixed dose of 10 mg per day
  Other Names: Lexapro
Drug: Bupropion XL — Fixed dose of 150 mg per day
  Other Names: Wellbutrin XL
  Arms: 2

SUMMARY:
This study will examine whether measures of brain electrical signals taken after a week of antidepressant medication treatment can predict whether a full treatment regimen will be effective.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common psychiatric illness with a high cost to society and individual patients. Initial medication treatments for MDD are often ineffective, precipitating a need to try other medications. This extends suffering, continues functional disability, and increases both the risk of relapse and the risk that people will abandon treatment. Having a biological marker of likely treatment effectiveness to predict and guide clinicians' decisions would reduce the likelihood of people with MDD experiencing unsuccessful treatments. This study will test whether quantitative electroencephalogram (QEEG) measures taken after 1 week of medication treatment can predict effectiveness of a full treatment regimen with depression medications.

Participation in this study will last 8 weeks. At the first study visit, participants will undergo baseline assessments. These assessments will include an interview about present condition, medical and psychiatric history, and past and current medication treatments; a urine test; and questionnaires about depression symptoms and other possible symptoms. The study doctor may ask for other assessments based on each participant's individual profile.

Participants will then complete a 1-week treatment with escitalopram, a type of antidepressant medication called a selective serotonin reuptake inhibitor (SSRI). At the first visit and again after the week-long escitalopram treatment, participants will undergo an electroencephalogram (EEG), which measures brain electrical activity. Based on certain measurements obtained from the EEG, an antidepressant treatment response (ATR) score will be calculated.

Participants will then be divided into two treatment groups: those who continue to receive escitalopram and those who begin treatment with bupropion XL, a non-SSRI antidepressant medication. Treatment for both groups will last 8 weeks, during which time participants will attend seven study visits. At these study visits, participants will be asked about how they are feeling, side effects, and benefit from the treatment. Further tests-such as a physical exam, lab test, or EEG-may be performed if study doctors think they are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for diagnosis of major depressive disorder (MDD) based on the Mini-International Neuropsychiatric Interview (MINI)
* Score greater than or equal to 12 on the Quick Inventory of Depressive Symptomatology - Self Rated version (QIDS-SR16)

Exclusion Criteria:

* Serious or unstable medical illness that would prevent complete participation in the trial, determined as needed from physical examination, electrocardiogram (ECG), laboratory safety tests, and review of systems
* Mentally or legally incapacitated and therefore unable to give informed consent
* Meets DSM-IV criteria for anorexia nervosa, bulimia nervosa, obsessive-compulsive disorder, any cognitive disorder, bipolar disorder, psychotic disorder, or major depression with psychotic features
* Diagnosis of a DSM-IV axis II disorder that would interfere with completion of the protocol
* Would have met criteria for a diagnosis of drug dependency or substance abuse within the preceding 9 months
* Stable and in remission on current psychotropic medication(s)
* Has had a course of electroconvulsive therapy (ECT) within the past 6 months
* Started psychotherapy for the current depressive episode within the past 2 months
* Has experienced treatment failure with an adequate trial of any study medication during the current episode of depression or has failed to tolerate escitalopram in the current episode
* Known contraindication for use of any of the study drugs, including hyponatremia during past use of a selective serotonin reuptake inhibitor (SSRI)
* Treated with fluoxetine or a monoamine oxidase inhibitor (MAOI) within the past 4 weeks
* Presence of a serious or unstable medical illness, including heart, liver, kidney, respiratory, endocrine, neurologic, or blood disease severe enough to significantly affect brain function or to interfere with interpretation of study results
* History of seizures, brain surgery, skull fracture, significant head trauma, or abnormal electroencephalogram (EEG)
* Currently pregnant or of childbearing potential and not using a medically acceptable means of birth control (e.g., oral contraceptive pill or implant, condom, diaphragm, spermicide, intrauterine device [IUD], past tubal ligation, partner with vasectomy)
* Breastfeeding
* University student or staff member directly under instruction, supervision, or employment of any of the investigators
* Requires hospitalization (e.g., poses an imminent danger to self or others)
* Initial quantitative EEG (QEEG) is contaminated with artifact so that determination of the biomarker is precluded
* Use of medications known to affect brain function

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Score on Hamilton Depression Rating Scale (HAM-D) | Measured nine times over 8 weeks

SECONDARY OUTCOMES:
Score on Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) | Measured nine times over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian A. Cook, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States